CLINICAL TRIAL: NCT06061224
Title: The Influences of Duration and Intensity of Early Mobilization on Myokines, Body Composition and Outcomes of Septic Patients in Intensive Care Unit
Brief Title: The Influences of Early Mobilization on Myokines, Body Composition and Outcomes in ICU Septic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202102342B0
Record Dates: First submitted 2023-09-05; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-08

CONDITIONS: Sepsis
Keywords: sepsis; early mobilization; myokines; body composition
MeSH Terms: conditions — Sepsis | interventions — Early Ambulation; Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non-PT group (No Intervention): with no physical treatment intervention (group 1)
- Early-PT group (Experimental): with physical treatment intervention started in ICU admission day 3 (group 2)
  Interventions: Behavioral: early mobilization (physical therapy)
- Delayed-PT (Experimental): with physical treatment intervention started after ICU admission day 3 (group 3)
  Interventions: Behavioral: early mobilization (physical therapy)

INTERVENTIONS:
Behavioral: early mobilization (physical therapy) — The investigators will consult rehabilitation department for Physical Therapy and patients will be grouped as clinically allocation.
  Protocols for consideration of initiation The timing is 72 hours after admission to ICU, early mobilization doses and duration is as the protocol of rehabilitation department
  Arms: Delayed-PT; Early-PT group

SUMMARY:
the investigators' preliminary data revealed that early physical therapy in patients with sepsis in ICU could promote recovery of function (liver and kidney) and decrease the length of stay in hospitalization. The levels of plasma IL-6 and IL-10 were higher in non-survival group than in survival group. the investigators hypothesize that myokines and body composition parameters are related to the prognosis of sepsis.the investigators will investigate the influences of duration and intensity of early mobilization on myokines, body composition and outcomes of septic patients in intensive care. The proposed study can help precision medicine in the future.

DETAILED DESCRIPTION:
The septic patients admitted to the intensive care unit (ICU) will be divided into three groups. One is non-PT group, with no physical treatment intervention (group 1), Early-PT group with physical treatment intervention started in ICU admission day 3 (group 2), and Delayed-PT with physical treatment intervention started after ICU admission day 3 (group 3). The grouping will be based on clinical indication for early mobilization (physical therapy) as below. The body composition data (of day 1, 3, 8) of the patients in the three groups will be measured, and the residual blood from day 1 and day 8 will be collected for detecting myokines.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aadmission in ICU 2. Clinical diagnosis of sepsis

Exclusion Criteria:

* 1. Expired in 3-days 2. Cardiac stents or pacemakers 3. Airborne disease 4. Contact-transmitted disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | The day discharged from ICU, "through study completion, an average of 1 year".
  Status of survival or mortality at the time discharged from ICU
Hospital mortality | The day discharged from hospital, "through study completion, an average of 1 year".
  Status of survival or mortality at the time discharged from hospital
7-day mortality | Day 7 after hospital admission
  Status of survival or mortality at Day 7 during hospital stay
28-day mortality | Day 28 after hospital admission
  Status of survival or mortality at Day 28 during hospital stay
90-day mortality | Day 90 after hospital admission
  Status of survival or mortality at Day 90 during hospital stay
ICU Days | During hospitalization, "through study completion, an average of 1 year".
  length of ICU stay
Change of white blood cell between day 1 and day 8 | Day 1 and Day8 after ICU admission
  assessing the change of white blood cell count between day 1 and day 8
Ventilation days | During hospitalization, "through study completion, an average of 1 year".
  Total using days of mechanical ventilation
Change of percentage of body fat between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of percentage of body fat between day 1 and day 8 by noninvasively Bio-electrical Impedance Analysis (BIA)
Change of total body water between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of total body water between day 1 and day 8 by noninvasively Bio-electrical Impedance Analysis (BIA)
Change of soft lean mass between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of soft lean mass between day 1 and day 8 by noninvasively Bio-electrical Impedance Analysis (BIA)
Concentration of serum IL-6 change between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of IL-6 between day 1 and day 8 by enzyme-linked immunosorbent assay (ELISA)
Concentration of serum BDNF change between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of serum BDNF between day 1 and day 8 by enzyme-linked immunosorbent assay (ELISA)
Concentration of serum IL-15 change between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of serum IL-15 between day 1 and day 8 by enzyme-linked immunosorbent assay (ELISA)
Concentration of serum SPARC change between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of serum SPARC (secreted protein acidic and rich in cysteine) between day 1 and day 8 by enzyme-linked immunosorbent assay (ELISA)
Concentration of serum Irisin change between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of serum Irisin between day 1 and day 8 by enzyme-linked immunosorbent assay (ELISA)
Concentration of serum Myostatin change between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of serum Myostatin between day 1 and day 8 by enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: FANG WEN-FENG, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan